CLINICAL TRIAL: NCT06033885
Title: Changes in User Satisfaction and Quality of Life Following 4 Weeks of Instrumented Standing Frame Intervention in Children With Disabilities - a Feasibility Intervention Study
Brief Title: User Satisfaction of an Instrumented Standing Frame
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: R82 A/S (Unknown); Innovation Fund Denmark (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11.928
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Functional Disability
Keywords: Children; Adolescents; Standing frame

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4-week control period + 4-week intervention period (Experimental): Prior to the intervention a 4-week control period, where the non-instrumented standing frame is used according to current practice, will be carried out. Subsequently, a 4-week intervention period, where the standing frame is instrumented (PONDUS®) allowing continued adjustments of the force and position within and between sessions will be conducted.
  Interventions: Device: PONDUS®

INTERVENTIONS:
Device: PONDUS® — PONDUS® is a CE-marked medical device to support the positioning of the user in a R82 standing frame.
  PONDUS® is designed as a pair of instrumented foot plates and an app as an external display.
  PONDUS® gives individual readings from the right and the left plate telling how much force is applied to each plate by combining high frequency data from three pressure sensors in each plate. The data is displayed in the app as a time series graph and can also be exported.

SUMMARY:
Standing frames have existed for a long time and are well-established medical devices used to allow weight bearing in standing for persons who are unable to stand independently.

Documenting the effectiveness of interventions using standing frames is complex. The current evidence base for their use is limited due to studies of low to moderate quality and small effects documented.

Providing real-time feed-back on force and position and thus continuous tracking of the intensity allows for informed decision making about the support provided by the standing frame in clinical settings, thereby making it possible to document the potential setup for optimal support and potential association between the intensity and positive effects of the standing frames.

The objective of the study is to document potential short-term benefits on a) patient satisfaction and health-related quality of life and b) changes in prescription from the prescribing therapist of the use of standing frames in children with standing disabilities when PONDUS®, a digital product used to assess the force applied during standing in a R82 standing frame is applied opposed to current practice.

The study is a one-arm feasibility intervention study using participants as their own controls. The study will include 15 children with functional disabilities who currently uses a standing frame.

DETAILED DESCRIPTION:
Most children stand independently by the age of 11 month, allowing them to apply different loads on their bones, joints, and muscles, and experience their surroundings from a new perspective. Children who do not reach the motor milestone "standing" in early childhood should have access to assistive medical devices such as standing frames, which enable them to gain benefits of the standing position as typically developing children.

Standing frames have existed for a long time and are well-established medical devices used to allow weight bearing in standing for persons who are unable to stand independently. The frame supports the child with upholstered plates and straps around the legs, trunk and/or head and is often positioned in an almost vertical posture, allowing the user partial weight bearing on their lower extremities. The devices are widely used as part of postural management for persons with disability and a population-based study in Sweden shows that 31% of all children with cerebral palsy use external support to stand.

Documenting the effectiveness of interventions using standing frames is complex. The current evidence base for their use is limited due to studies of low to moderate quality and small effects documented. A systematic review and recent studies on the potential benefits of using standing frames indicate improvements in a range of functions and activities including: mental functions, bone and joint development and health, cardiovascular and respiratory systems, digestive systems and urinary functions, neuromusculoskeletal and movement related functions, pain, mobility, the ability to maintain a sitting or standing position, and major life areas, including interaction with peers. Importantly, the studies did not report adverse events or serious harm.

The above studies reveal a large variety in dosing in terms of frequency and time of use of the standing frames from <1 to 7 days per week, 1 or more sessions per day and <30 min to >120 min per session. Importantly, none of the studies document dosing in terms of intensity assessed as the degree of weight bearing while using a standing frame. Multiple variables such as type of frame, use of supports, inclination, activities performed while standing and inclination of the frame have been suggested to affect weight bearing in standing frames. Instrumented standing frames have been used in experimental settings and have documented a large variation in percentage of body weight from 23-133%, which could indicate serious issues of controlling the intensity or even misuse and/or measurement error. To our knowledge, instrumented standing frames that can assess force and position during the use of a standing frames is currently not available for use in clinical practice.

The lack of information about force and position during the use of standing frames in clinical settings makes it impossible to document the potential setup for optimal support and potential association between the intensity and positive effects of the standing frames and, moreover, whether the intensity of the intervention should be tailored to the individual child.

Providing real-time feed-back on force and position and thus continuous tracking of the intensity allows for informed decision making about the support provided by the standing frame in a clinical setting.

The purpose of this study is to document potential short-term benefits on a) patient satisfaction and health-related quality of life and b) changes in prescription from the prescribing therapist of the use of standing frames in children with standing disabilities when PONDUS®, a digital product used to assess the force applied during standing in a R82 standing frame, is applied opposed to current practice.

The study is a one-arm feasibility intervention study using participants as their own controls. The study will be conducted in special day-care centers and schools or in the children's home. Participants will be 15 children with functional disabilities in the age of 3-17 years who currently uses a standing frame.

Recruitment will be conducted in collaboration with the study's commercial partner's distributor network and special day-care centers and schools across Denmark, that will assist in identifying possible study participants. In addition to the above parents will be reached through advocacy organizations or on social medias with an invitation for participation in the studies.

Prior to the intervention a 4-week control period, where the non-instrumented standing frame is used according to standard practice, will be carried out. Subsequently, a 4-week intervention period, where the standing frame is instrumented (PONDUS®) allowing continued monitoring and adjustments of the force and position during sessions will be conducted. Changes in outcome measures will be evaluated as the difference in within-group change score between the control period and intervention period.

Participation in the study will be voluntary and all participants will be informed that even after the eventual acceptance of participation, at any stage of the project they may decide to discontinue participation in the trial without giving any reason and without it having consequences for further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children with disabilities aged 3-17 years who uses a standing frame
* Informed consent from parents
* Informed consent from children aged 15-17 years

Exclusion Criteria:

* Earlier interventions in the form of orthopedic surgery within the past 52 weeks
* Injections with botulinum toxin type A in the 12 weeks prior to baseline assessments
* Insufficient co-operation and cognitive understanding to participate in the study
* Planned interventions in form of orthopedic surgery and/or botulinum toxin type A in the study period

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with an instrumented standing frame | 8 weeks difference in change score between the control period and intervention period
  Patient satisfaction with an instrumented standing frame will be assessed with the Quebec User Evaluation of Satisfaction with Assistive Technology (Quest 2.0) questionnaires eight items assessing characteristics of the assistive device in terms of the following dimensions: 1) dimensions (size), 2. weight, 3. adjustments, 4. safety, 5. durability, 6. simplicity of use, 7. comfort and 8. effectiveness.
  For each item, the questionnaire uses a 5point scale, 1 being not satisfied at all and 5 being very satisfied.

SECONDARY OUTCOMES:
The three most important aspects of patient satisfaction with an instrumented standing frame | 8 weeks difference in change score between the control period and intervention period
  Through user involvement, the three key aspects of patient satisfaction with an instrumented standing frame will be selected from the Quebec User Evaluation of Satisfaction with Assistive Technology (Quest 2.0) questionnaire
Usability of an instrumented standing frame | 8 weeks difference in change score between the control period and intervention period
  Usability of an instrumented standing frame will be assessed with the Usefulness, Satisfaction, and Ease of use (USE) Questionnaire.
  For each item, the questionnaire uses a 7 point Likert rating scales, with 1 = Strongly disagree to 7 = Strongly agree.
Health-related quality of life | 8 weeks difference in change score between the control period and intervention period
  Health-related quality of life will be assessed with the Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) questionnaire.
  Scores for each domain and for the total survey are standardized and range from 0 (worse) to 100 (best).
Changes in prescription from the prescribing therapist | 8 weeks difference in change score between the control period and intervention period
  Changes in prescription from the prescribing therapist of the use of the standing frame when PONDUS® is applied opposed to current practice will be assessed with a self-constructed questionnaire made for the purpose

OTHER OUTCOMES:
Patient satisfaction with assistive device service of an instrumented standing frame | 8 weeks difference in change score between the control period and intervention period
  Patient satisfaction with assistive device service of an instrumented standing frame will be assessed with the Quebec User Evaluation of Satisfaction with Assistive Technology (Quest 2.0) questionnaires four items assessing characteristics of service in terms of the following dimensions: 1. service delivery, 2. repairs and service of the device, 3. professionalism of service and 4. follow-up service.
  For each item, the questionnaire uses a 5point scale, 1 being not satisfied at all and 5 being very satisfied.
Patient satisfaction with PONDUS® | 4 weeks score from the intervention period
  Patient satisfaction with PONDUS® will be assessed with the Quebec User Evaluation of Satisfaction with Assistive Technology (Quest 2.0) questionnaire.
  For each item, the questionnaire uses a 5point scale, 1 being not satisfied at all and 5 being very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Holsgaard-Larsen, Professor, Principal Investigator — Department of Clinical Research, SDU & Department of Orthopaedics and Traumatology, OUH
Locations (1):
- University of Southern Denmark, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to ethical and legal considerations, our data cannot be shared publicly. This is due to the restrictions from the Regional and the National Committee on Health Research Ethics and the General Data Protection Regulation (EU) 2016/679, since the data contains person-specific information on birth date, sex, and diagnosis classification among other.
  Data are available for researchers who meet the criteria for access to confidential data. Access may be acquired through contact to the research group.

REFERENCES:
- [Background] WHO Multicentre Growth Reference Study Group. WHO Motor Development Study: windows of achievement for six gross motor development milestones. Acta Paediatr Suppl. 2006 Apr;450:86-95. doi: 10.1111/j.1651-2227.2006.tb02379.x. PMID 16817682
- [Background] Wijnhoven TM, de Onis M, Onyango AW, Wang T, Bjoerneboe GE, Bhandari N, Lartey A, al Rashidi B. Assessment of gross motor development in the WHO Multicentre Growth Reference Study. Food Nutr Bull. 2004 Mar;25(1 Suppl):S37-45. doi: 10.1177/15648265040251S105. PMID 15069918
- [Background] Goodwin J, Lecouturier J, Smith J, Crombie S, Basu A, Parr JR, Howel D, McColl E, Roberts A, Miller K, Cadwgan J. Understanding frames: A qualitative exploration of standing frame use for young people with cerebral palsy in educational settings. Child Care Health Dev. 2019 May;45(3):433-439. doi: 10.1111/cch.12659. PMID 30883842
- [Background] Paleg GS, Smith BA, Glickman LB. Systematic review and evidence-based clinical recommendations for dosing of pediatric supported standing programs. Pediatr Phys Ther. 2013 Fall;25(3):232-47. doi: 10.1097/PEP.0b013e318299d5e7. PMID 23797394
- [Background] Rodby-Bousquet E, Hagglund G. Sitting and standing performance in a total population of children with cerebral palsy: a cross-sectional study. BMC Musculoskelet Disord. 2010 Jun 23;11:131. doi: 10.1186/1471-2474-11-131. PMID 20573201
- [Background] Rivi E, Filippi M, Fornasari E, Mascia MT, Ferrari A, Costi S. Effectiveness of standing frame on constipation in children with cerebral palsy: a single-subject study. Occup Ther Int. 2014 Sep;21(3):115-23. doi: 10.1002/oti.1370. Epub 2014 May 16. PMID 24838311
- [Background] Capati V, Covert SY, Paleg G. Stander Use for an Adolescent with Cerebral Palsy at GMFCS Level with Hip and Knee Contractures. Assist Technol. 2020 Nov 1;32(6):335-341. doi: 10.1080/10400435.2019.1579268. Epub 2019 Apr 4. PMID 30945990
- [Background] Han EY, Choi JH, Kim SH, Im SH. The effect of weight bearing on bone mineral density and bone growth in children with cerebral palsy: A randomized controlled preliminary trial. Medicine (Baltimore). 2017 Mar;96(10):e5896. doi: 10.1097/MD.0000000000005896. PMID 28272197
- [Background] Macias-Merlo L, Bagur-Calafat C, Girabent-Farres M, A Stuberg W. Effects of the standing program with hip abduction on hip acetabular development in children with spastic diplegia cerebral palsy. Disabil Rehabil. 2016;38(11):1075-81. doi: 10.3109/09638288.2015.1100221. Epub 2015 Oct 30. PMID 26517269
- [Background] Macias-Merlo L, Bagur-Calafat C, Girabent-Farres M, Stuberg WA. Standing Programs to Promote Hip Flexibility in Children With Spastic Diplegic Cerebral Palsy. Pediatr Phys Ther. 2015 Fall;27(3):243-9. doi: 10.1097/PEP.0000000000000150. PMID 26020594
- [Background] Hough JP, Boyd RN, Keating JL. Systematic review of interventions for low bone mineral density in children with cerebral palsy. Pediatrics. 2010 Mar;125(3):e670-8. doi: 10.1542/peds.2009-0292. Epub 2010 Feb 1. PMID 20123765
- [Background] Salem Y, Lovelace-Chandler V, Zabel RJ, McMillan AG. Effects of prolonged standing on gait in children with spastic cerebral palsy. Phys Occup Ther Pediatr. 2010 Feb;30(1):54-65. doi: 10.3109/01942630903297177. PMID 20170432
- [Background] Curtis DJ, Woollacott M, Bencke J, Lauridsen HB, Saavedra S, Bandholm T, Sonne-Holm S. The functional effect of segmental trunk and head control training in moderate-to-severe cerebral palsy: A randomized controlled trial. Dev Neurorehabil. 2018 Feb;21(2):91-100. doi: 10.1080/17518423.2016.1265603. Epub 2017 Jan 3. PMID 28045553
- [Background] Curtis DJ, Butler P, Saavedra S, Bencke J, Kallemose T, Sonne-Holm S, Woollacott M. The central role of trunk control in the gross motor function of children with cerebral palsy: a retrospective cross-sectional study. Dev Med Child Neurol. 2015 Apr;57(4):351-7. doi: 10.1111/dmcn.12641. Epub 2014 Nov 20. PMID 25412902
- [Background] Pedlow K, McDonough S, Lennon S, Kerr C, Bradbury I. Assisted standing for Duchenne muscular dystrophy. Cochrane Database Syst Rev. 2019 Oct 13;10(10):CD011550. doi: 10.1002/14651858.CD011550.pub2. PMID 31606891
- [Background] Paleg G, Altizer W, Malone R, Ballard K, Kreger A. Inclination, hip abduction, orientation, and tone affect weight-bearing in standing devices. J Pediatr Rehabil Med. 2021;14(3):433-441. doi: 10.3233/PRM-190660. PMID 34057103
- [Background] Herman D, May R, Vogel L, Johnson J, Henderson RC. Quantifying weight-bearing by children with cerebral palsy while in passive standers. Pediatr Phys Ther. 2007 Winter;19(4):283-7. doi: 10.1097/PEP.0b013e318156cc4d. PMID 18004195
- [Background] Kecskemethy HH, Herman D, May R, Paul K, Bachrach SJ, Henderson RC. Quantifying weight bearing while in passive standers and a comparison of standers. Dev Med Child Neurol. 2008 Jul;50(7):520-3. doi: 10.1111/j.1469-8749.2008.03021.x. PMID 18611202